CLINICAL TRIAL: NCT05982496
Title: 18F-FES PET/MRI for Tailoring Treatment of Luminal a and Lobular Breast Cancer: a Phase II Prospective Cohort Study Evaluating the Performance of FES PET/MRI in Axillary Staging Compared with Axillary Surgery
Brief Title: 18F FES-PET/MRI for Tailoring Treatment of Luminal a and Lobular Breast Cancer
Acronym: FESTA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Rosa Di Micco, MD, Principal Investigator, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FESTA
Record Dates: First submitted 2023-07-05; First posted 2023-08-08 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Female; Lobular Breast Carcinoma; PET/MRI; Axillary Lymphadenopathy; Luminal a Breast Cancer
MeSH Terms: conditions — Carcinoma, Lobular

STUDY DESIGN:
Intervention Model Description: Cohort A
  * candidates to surgery as first treatment regardless of cN
  * ER+ Her2 negative BC with ki67>10% Cohort B
  * ER positive BC treated with induction ET Cohort C
  * candidates to neoadjuvant chemotherapy Cohort D
  * Metastatic LumA or ER-positive Lob BC, at first diagnosis or in progression
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A (Experimental): * Candidates to surgery as first treatment regardless of cN
  * ER+ Her2 negative BC with ki67>10%
  Interventions: Drug: FES; Procedure: PET/MRI A; Genetic: Translational analysis
- Cohort B (Experimental): • ER positive BC treated with induction ET
  Interventions: Drug: FES; Procedure: PET/MRI B; Genetic: Translational analysis
- Cohort C (Experimental): • Candidates to neoadjuvant chemotherapy
  Interventions: Drug: FES; Procedure: PET/MRI C; Genetic: Translational analysis
- Cohort D (Experimental): • Metastatic LumA or ER-positive Lob BC, at first diagnosis or in progression
  Interventions: Drug: FES; Procedure: PET/MRI D; Genetic: Translational analysis

INTERVENTIONS:
Drug: FES — 16-alpha-18F-fluoro-17-beta-estradiol(FES) is a radiolabeled form of estrogen binding to functionally active ER which will be used as radiotracer for the PET/MRI exam
Procedure: PET/MRI A — An additional FES PET/MRI will be performed before surgery.
  Arms: Cohort A
Procedure: PET/MRI B — Two additional PET/MRI will be performed before and after induction ET.
  Arms: Cohort B
Procedure: PET/MRI C — Two additional PET/MRI will be performed before and after two cycles of neoadjuvant chemotherapy.
  Arms: Cohort C
Procedure: PET/MRI D — Two additional PET/MRI will be performed before and after two cycles of systemic therapy.
  Arms: Cohort D
Genetic: Translational analysis — Selected cases of heterogeneous tumors on imaging will be also investigated on pathology, imaging, genomic and radiomic levels.

SUMMARY:
Study hypothesis is that combining the advantages of hybrid PET/MRI and the high sensitivity/specificity of 16-alpha-18F-fluoro-17-beta-estradiol(FES), a radiolabeled form of estrogen binding to functionally active ER, the investigators could obtain a reliable, non-invasive, operator-independent, one-stage imaging method for staging LumA and ER-positive Lobular tumours.

DETAILED DESCRIPTION:
This is a single-centre prospective cohort study where patients with LumA and ER-positive Lob will be enrolled in 4 cohorts undergoing: primary surgery; induction endocrine therapy; neoadjuvant chemotherapy; systemic therapy for metastatic disease. For the purpose of the study an additional FES PET/MRI exam will be performed at baseline for local and systemic staging and a second exam after systemic therapy. Correlations between FES PET/MRI parameters and pathology, gene expression and FDG PET parameters, when available, will be investigated. Aim 1: Evaluating the performance of FES PET/MRI in axillary staging compared with axillary surgery. Aim 2: Evaluating potential correlations between changes in FES uptake and changes in proliferation index after 3 weeks of endocrine therapy before surgery. Aim 3: Evaluating the performance of FES PET/MRI in staging of patients undergoing systemic therapy in comparison with standard imaging. Additionally, biological determinants of tumor heterogeneity will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age>= 18 yrs, diagnosed with primary or advanced breast cancer
* LumA or ER-positive Lobular subtypes Cohort A

  * candidates to surgery as first treatment regardless of cN
  * ER-positive Her2 negative BC with ki67>10% Cohort B
  * ER positive BC treated with induction ET Cohort C
  * candidates to neoadjuvant chemotherapy Cohort D
  * Metastatic LumA or ER-positive Lob BC, at first diagnosis or in progression

Exclusion Criteria:

* ER-negative tumors
* Pregnancy;
* Contraindication to PET;
* Contraindication to MRI;
* Claustrophobia;
* Allergy to the MR contrast agent;
* Severe renal insufficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of FES PET/MRI in detecting macrometastatic axillary lymph nodes | Day 50
  Ability of FES PET/MRI to detect macrometastatic (tumor deposit>2mm) axillary lymph nodes in BC patients with LumA or Lob who are candidates to primary surgery.

SECONDARY OUTCOMES:
Changes in Standard Uptake Value (SUV) of FES in patients undergoing induction Endocrine Treatment (ET) | Day 0 and Day 50
  To investigate the potential correlation between Δ(FES SUV) and Δ(Ki-67 as proliferation index) after induction ET in luminal BC.

OTHER OUTCOMES:
FES PET/MRI sensitivity compared to that of standard imaging in patients undergoimg systemic therapy for neoadjuvant purposes or for metastatic disease. | Day 0
  Results from FES PET/MRI will be compared with those from standard imaging in terms of sensitivity and number of lesions detected.
FES PET/MRI ability to predict tumor response or no response to therapy | Day 180
  Results of FES PET/MRI after two cycles of therapy will be compared to final pathology (cohort C) or standard imaging at 6 months (cohort D)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franquet E, Park H. Molecular imaging in oncology: Common PET/CT radiopharmaceuticals and applications. Eur J Radiol Open. 2022 Nov 24;9:100455. doi: 10.1016/j.ejro.2022.100455. eCollection 2022. PMID 36439301
- [Background] Schumacher K, Inciardi M, O'Neil M, Wagner JL, Shah I, Amin AL, Balanoff CR, Larson KE. Is axillary imaging for invasive lobular carcinoma accurate in determining clinical node staging? Breast Cancer Res Treat. 2021 Feb;185(3):567-572. doi: 10.1007/s10549-020-06047-w. Epub 2021 Jan 3. PMID 33389408
- [Background] Iorfida M, Maiorano E, Orvieto E, Maisonneuve P, Bottiglieri L, Rotmensz N, Montagna E, Dellapasqua S, Veronesi P, Galimberti V, Luini A, Goldhirsch A, Colleoni M, Viale G. Invasive lobular breast cancer: subtypes and outcome. Breast Cancer Res Treat. 2012 Jun;133(2):713-23. doi: 10.1007/s10549-012-2002-z. Epub 2012 Mar 8. PMID 22399188